CLINICAL TRIAL: NCT06340568
Title: A Phase III, Randomized, Multi-site, Open-label Trial of BNT323/DB-1303 Versus Investigator's Choice of Chemotherapy in Previously Treated Patients With HER2- Expressing Recurrent Endometrial Cancer
Brief Title: A Clinical Study of the Anti-cancer Effects of an Investigational Therapy or Chemotherapy in Patients With Recurring Uterine Cancer
Acronym: Fern-EC-01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: DualityBio Inc. (Industry); BioNTech (Shanghai) Pharmaceuticals Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT323-01; GOG-3105 (Other: Gynecologic Oncology Group Foundation); 2023-507525-42-00 (EU CTIS Number); ENGOT- EN25/NSGO-CTU (Other: European Network for Gynaecological Oncological Trial and Nordic Society of Gynaecological Oncology Clinical Trial Unit)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
Keywords: Human epidermal growth factor receptor 2 (HER2); HER2-expressing tumors; Recurrent endometrial cancer; IHC scores 1+, 2+, and 3+; Immune checkpoint inhibitor; Platinum-based therapy; HER2 protein expression; HER2-expressing endometrial cancer; ErbB-2 receptor; Antibody drug conjugate (ADC)
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Doxorubicin; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (HER2 IHC score 1+ or 2+): BNT323/DB-1303 (Experimental)
  Interventions: Drug: BNT323/DB-1303
- Cohort 1 - Doxorubicin or paclitaxel (or docetaxel) (Active Comparator): Single agent chemotherapy (either doxorubicin or paclitaxel) per investigator's choice. Participants with contraindications to paclitaxel may receive docetaxel as an alternative (if available at the site).
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel; Drug: Docetaxel
- Cohort 2 (HER2 IHC score 3+) - BNT323/DB-1303 (Experimental)
  Interventions: Drug: BNT323/DB-1303

INTERVENTIONS:
Drug: BNT323/DB-1303 — intravenous (IV) infusion
  Other Names: trastuzumab pamirtecan
  Arms: Cohort 1 (HER2 IHC score 1+ or 2+): BNT323/DB-1303; Cohort 2 (HER2 IHC score 3+) - BNT323/DB-1303
Drug: Doxorubicin — IV bolus or infusion
  Arms: Cohort 1 - Doxorubicin or paclitaxel (or docetaxel)
Drug: Paclitaxel — IV infusion
  Arms: Cohort 1 - Doxorubicin or paclitaxel (or docetaxel)
Drug: Docetaxel — IV infusion
  Arms: Cohort 1 - Doxorubicin or paclitaxel (or docetaxel)

SUMMARY:
The study is divided into two cohorts (Cohort 1 and Cohort 2), to which participants will be enrolled based on the amount of human epidermal growth factor receptor 2 (HER2) in their tumor sample.

In Cohort 1, the main goal is to assess how well BNT323 (also known as DB-1303) or chemotherapy (doxorubicin or paclitaxel [or docetaxel, if participants cannot take paclitaxel]) works by determining the progression-free survival (PFS) of participants who have been previously treated with immune checkpoint inhibitors (ICIs).

In Cohort 2, the main goal is to assess how well BNT323 works by determining the objective response rate (ORR), that is, the percentage of participants whose tumor shrinks (partial response) or disappears (complete response) after treatment.

The safety of BNT323 will also be assessed by following the occurrence of unfavorable/adverse effects that are seen after treatment. Other measures include the pharmacokinetics of BNT323 (or how BNT323 moves through and out of the body), the body's immune response, and the impact on quality of life.

DETAILED DESCRIPTION:
This is an open-label, randomized, multi-site, Phase III, interventional clinical study designed to determine the efficacy and safety of BNT323 compared with investigator's choice of single agent chemotherapy in previously treated participants with recurrent endometrial cancer (including HER2 1+ or 2+ score as determined using a centralized immunohistochemistry [IHC] analysis method), whose disease has progressed on at least one line of platinum-based therapy and ICI (Cohort 1). In addition, participants with recurrent endometrial cancer with HER2 IHC 3+ score will be enrolled in a BNT323 monotherapy arm (Cohort 2) to further investigate the efficacy and safety of BNT323.

In Cohort 1, participants will be randomized 2:1 to receive either BNT323/DB-1303 or investigator's choice of single agent chemotherapy, preferably doxorubicin or paclitaxel (or docetaxel if contraindicated to paclitaxel and available at the site) until Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) defined progressive disease (PD) unless there is unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation is met.

In Cohort 2, participants will receive BNT323 monotherapy until RECIST v1.1 defined PD unless there is unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation is met.

The study consists of a screening period, a treatment period, a safety follow-up period, an efficacy follow-up period, and a long-term survival follow-up. The expected treatment duration per participant is ~6 months, followed by an anticipated long-term survival follow-up period of up to 53 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Are female adults (defined as ≥18 years of age or acceptable age according to local regulations at the time of voluntarily giving informed consent).
* Have histologically confirmed endometrial cancer that:

  * Is recurrent,
  * Has a HER2 IHC score of 1+, 2+ (Cohort 1), or 3+ (Cohort 2) as determined by central laboratory testing for HER2 expression, and
  * Is not defined as a true sarcoma (i.e., leiomyosarcoma or endometrial stromal sarcoma). Note: Uterine carcinosarcoma is allowed.
* Have measurable disease defined by RECIST v1.1.
* Have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
* Have recurrent endometrial cancer and meet any of the following:

  * developed recurrence <12 months from completing platinum-based chemotherapy given as adjuvant therapy for Stage I to III disease, or
  * developed recurrence after platinum-based chemotherapy in the recurrent/metastatic setting.
* Have received prior ICI treatment (i.e., anti-programmed death 1/anti-programmed death-ligand 1)
* Have a life expectancy of ≥12 weeks at screening.

Key Exclusion Criteria:

* Are ineligible for all options in the investigator's choice of chemotherapy arm, per local prescribing information and institutional guidelines (applicable to Cohort 1 only).
* Have a history of small bowel obstruction requiring hospitalization within the past 3 months prior the first dose of study treatment.
* Have an uncontrolled intercurrent illness that would limit compliance with study requirement or substantially increase risk of incurring adverse events.
* Have clinically uncontrolled pleural effusion, ascites or pericardial effusion requiring drainage, or peritoneal shunt within 2 weeks prior to the first dose of study treatment.
* Have a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, have current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Participants with prior use of immunosuppressive medication within 14 days prior to the first dose of study treatment, except for intranasal and inhaled corticosteroids or systemic corticosteroids at doses of less than 10 mg/day of prednisone or equivalent, and topical corticosteroids. Participants receiving corticosteroids may continue if the dose is stable upon giving main informed consent.
* Have a lung-specific intercurrent clinically significant illness including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary emboli within 3 months prior to the first dose of study treatment, severe asthma, chronic obstructive pulmonary disorder with moderate acute exacerbations, restrictive lung disease, pulmonary fibrosis, radiation pneumonitis, significant pleural effusion etc.), or any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement (i.e., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis etc.), and/or prior pneumonectomy (complete).
* Have uncontrolled infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks prior to the first dose of study treatment.
* Have unresolved toxicities from previous anti-cancer therapy, defined as toxicities (other than alopecia, fatigue, or endocrinopathies that are well controlled) not yet resolved to Grade ≤1 or baseline.
* Are pregnant or breastfeeding or are planning pregnancy during the study or within 7 months after the last dose of study treatment.
* Have a history of allergies, hypersensitivities, or intolerance to study treatments (investigational medicinal products and auxiliary medicinal product) including any excipients thereof or to other monoclonal antibodies. Participants who have successfully undergone a desensitization process and are able to tolerate the drug are eligible.
* Had prior treatment with topoisomerase I inhibitors, including ADCs.
* Have left ventricular ejection fraction <55% by either echocardiography or multiple-gated acquisition within 28 days prior to the first dose of study treatment. This includes participants with tissue doppler E/e' ratio >15.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: PFS assessed by blinded independent central review (BICR) in participants with HER2 IHC 1+/2+ recurrent endometrial cancer | Up to approximately 53 months
  By treatment arm. Defined as the time from randomization to the first objective tumor progression (per RECIST v1.1) or death from any cause, whichever occurs first.
Cohort 2: ORR assessed by BICR in participants with HER2 IHC 3+ recurrent endometrial cancer | Up to approximately 53 months
  Defined as the proportion of participants with a CR or PR (per RECIST v1.1) as best overall response with confirmation.

SECONDARY OUTCOMES:
Cohort 1: Overall survival (OS) in participants with HER2 IHC 1+/2+ recurrent endometrial cancer | Up to approximately 53 months
  By treatment arm. Defined as the time from randomization to death from any cause.
Cohort 1: PFS assessed by the investigator in participants with HER2 IHC 1+/2+ recurrent endometrial cancer | Up to approximately 53 months
  By treatment arm. Defined as the time from randomization to the first objective tumor progression (per RECIST v1.1) or death from any cause, whichever occurs first.
Cohort 1: ORR assessed by BICR in participants with HER2 IHC 1+/2+ recurrent endometrial cancer | Up to approximately 53 months
  By treatment arm. Defined as the proportion of participants with a CR or PR (per RECIST v1.1) as best overall response with confirmation.
Cohort 1: ORR assessed by the investigator in participants with HER2 IHC 1+/2+ recurrent endometrial cancer | Up to approximately 53 months
  By treatment arm. Defined as the proportion of participants with a CR or PR (per RECIST v1.1) as best overall response with confirmation.
Cohort 1: Duration of response (DoR) assessed by BICR in participants with HER2 IHC 1+/2+ recurrent endometrial cancer | Up to approximately 53 months
  By treatment arm. Defined as the time from first objective response (CR or PR per RECIST v1.1) to first occurrence of objective tumor progression (PD per RECIST v1.1) or death from any cause, whichever occurs first.
Cohort 1: DoR assessed by the investigator in participants with HER2 IHC 1+/2+ recurrent endometrial cancer | Up to approximately 53 months
  By treatment arm. Defined as the time from first objective response (CR or PR per RECIST v1.1) to first occurrence of objective tumor progression (PD per RECIST v1.1) or death from any cause, whichever occurs first.
Cohort 1: Percentage of participants with HER2 IHC 1+/2+ recurrent endometrial cancer with occurrence of treatment-emergent adverse events (TEAEs) | Up to 35 days after the last dose of study treatment
  By treatment arm. TEAEs including Grade ≥3, serious, and fatal TEAEs by relationship.
Cohort 1: Percentage of participants with HER2 IHC 1+/2+ recurrent endometrial cancer with occurrence of TEAEs leading to drug interruption, dose reduction, or discontinuation of study treatment. | Up to 35 days after the last dose of study treatment
  By treatment arm.
Cohort 2: ORR assessed by the investigator participants with HER2 IHC 3+ recurrent endometrial cancer | Up to approximately 53 months
  Defined as the proportion of participants in whom a CR or PR (per RECIST v1.1) is observed as best overall response with confirmation.
Cohort 2: DoR assessed by BICR in participants with HER2 IHC 3+ recurrent endometrial cancer | Up to approximately 53 months
  Defined as the time from first objective response (CR or PR per RECIST v1.1) to first occurrence of objective tumor progression (PD per RECIST v1.1) or death from any cause, whichever occurs first.
Cohort 2: DoR assessed by the investigator in participants with HER2 IHC 3+ recurrent endometrial cancer | Up to approximately 53 months
  Defined as the time from first objective response (CR or PR per RECIST v1.1) to first occurrence of objective tumor progression (PD per RECIST v1.1) or death from any cause, whichever occurs first.
Cohort 2: PFS assessed by BICR in participants with HER2 IHC 3+ recurrent endometrial cancer | Up to approximately 53 months
  Defined as the time from the first dose of study treatment to the first objective tumor progression (per RECIST v1.1) or death from any cause, whichever occurs first.
Cohort 2: PFS assessed by the investigator in participants with HER2 IHC 3+ recurrent endometrial cancer | Up to approximately 53 months
  Defined as the time from the first dose of study treatment to the first objective tumor progression (per RECIST v1.1) or death from any cause, whichever occurs first.
Cohort 2: OS in participants with HER2 IHC 3+ recurrent endometrial cancer | Up to approximately 53 months
  Defined as the time from the first dose of trial treatment to death from any cause.
Cohort 2: Percentage of participants with HER2 IHC 3+ recurrent endometrial cancer with occurrence of TEAEs | Up to 35 days after the last dose of study treatment
  BNT323 monotherapy. TEAEs including Grade ≥3, serious, and fatal TEAEs by relationship.
Cohort 2: Percentage of participants with HER2 IHC 3+ recurrent endometrial cancer with occurrence of TEAEs leading to drug interruption, dose reduction, or discontinuation of study treatment. | Up to 35 days after the last dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (80):
- United States (3):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - The Center of Hope Reno, Reno, Nevada
  - Miami Valley Hospital South, Centerville, Ohio
- Argentina (4):
  - Hospital Británico de Buenos Aires, Buenos Aires
  - Investigaciones CORI S.R.L., La Rioja
  - Hospital Provincial del Centenario, Rosario
  - Centro Oncológico de Excelencia, San Juan
- Australia (7):
  - Adelaide Oncology & Haematology, Adelaide
  - Cancer Research SA, Adelaide
  - Gosford Hospital, Gosford
  - Frankston Hospital, Melbourne
  - Sunshine Hospital, Saint Albans
  - Mater Hospital Brisbane, South Brisbane
  - Wollongong Hospital, Wollongong
- Belgium (2):
  - UZ Leuven, Leuven
  - CHU UCL Namur-Sainte-Elisabeth, Namur
- Brazil (2):
  - Hospital de Clínicas de Passo Fundo, Passo Fundo
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
- Canada (3):
  - Jewish General Hospital, Montreal
  - Health Sciences Centre, St. John's
  - Princess Margaret Cancer C, Toronto
- China (25):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Gansu Provincial Maternity and Child-care Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
- Denmark (2):
  - Aalborg Universit Hospital, Aalborg
  - Rigshospitalet, Copenhagen
- France (3):
  - ICO - Site Paul Papin, Angers
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - Institut de Cancérologie de Strasbourg Europe - ICANS, Strasbourg
- Radboud UMC, Nijmegen, Netherlands
- South Korea (11):
  - Keimyung Univty Dongsan Hospital, Daegu
  - National Cancer Center, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
- Taiwan (6):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Kuang Tien General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - MacKay Memorial Hospital_ Taipei Branch, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (11):
  - Royal Sussex County Hospital, Brighton
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Castle Hill Hospital, Cottingham
  - Western General Hospital, Edinburgh
  - Royal Devon & Exeter HPT, Exeter
  - University College London Hospitals, London
  - Mount Vermont Cancer Center, Middlesex
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Singleton Hospital, Swansea
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Secord AA, Powell MA, McAlpine J. Molecular Characterization and Clinical Implications of Endometrial Cancer. Obstet Gynecol. 2025 Nov 1;146(5):660-671. doi: 10.1097/AOG.0000000000006080. Epub 2025 Sep 18. PMID 40966692